CLINICAL TRIAL: NCT04181450
Title: Biodex Balance System Cut-off Scores in Geriatric Individuals With Non-Specific Low Back Pain
Brief Title: Biodex Balance System Cut-off Scores in Geriatric Individuals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Principal Investigator, Hacettepe University
Other Study IDs: 2019800
Record Dates: First submitted 2019-11-25; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Low Back Pain; Balance; Distorted
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determination of the Cut-off Scores of Biodex Balance System — Based on the findings of the Sherafat et al. (Sherafat, S., Salavati, M., Takamjani, I. E., Akhbari, B., Mohammadirad, S., Mazaheri, M., & Negahban, H. (2013). Intrasession and intersession reliability of postural control in participants with and without nonspecific low back pain using the Biodex Balance System. Journal of manipulative and physiological therapeutics, 36(2), 111-118.) related to intrasession and intersession reliability of BBS in patients with NSLBP12, in the present study, one stability level (Level 5; ICC ≥0.70) and two conditions (eyes-open and eyes-closed) will be selected as testing procedure. All postural assessments will be performed during bilateral stance for a period of 30 seconds.

SUMMARY:
Low back pain (LBP) is an important musculoskeletal problem that causes clinical, social and economic losses. LBP, which affects approximately 85% of the lifetime population, becomes chronic LBP in 23% of individuals lasting 3 months or more. Although there are various forms of LBP, the most common form is non-specific low back pain (NSLBP). There are no specific and definable pathologies in NSLBP such as a history of spinal surgery, presence of neurological deficit, facet joint problem, disc herniation and sacroiliac joint dysfunction.

Biodex Balance System (Biodex Medical Systems, Shirley, NY) (BBS) is a device used for objective evaluation of static and dynamic balance, allowing free movement in mediolateral and anteroposterior directions. The validity-reliability studies of the BBS were conducted in various populations including active, non-active, young adult and geriatric individuals, and individuals with ankle sprains. The validity-reliability study of individuals with NSLBP was reported by Sherafat et al. has a strong-excellent correlation with four-square step test, timed-up-and-go test, Berg Balance Scale, and single leg stance test.

Studies have emphasized the use of BBS in geriatric individuals with NSLBP, but no data on the cut-off scores of this system have been found. The determination of a cut-off score with high sensitivity and specificity is thought to be beneficial for detecting deterioration in functional status in geriatric individuals with NSLBP. Therefore, the aim of our study is to determine BBS cut-off scores in geriatric individuals with NSLBP.

DETAILED DESCRIPTION:
Low back pain (LBP) is an important musculoskeletal problem that causes clinical, social and economic losses. LBP, which affects approximately 85% of the lifetime population, becomes chronic LBP in 23% of individuals lasting 3 months or more. Although there are various forms of LBP, the most common form is non-specific low back pain (NSLBP). There are no specific and definable pathologies in NSLBP such as a history of spinal surgery, presence of neurological deficit, facet joint problem, disc herniation and sacroiliac joint dysfunction.

Although there are studies examining the changes in various positions in geriatric individuals with NSLBP, maintaining and maintaining postural control during standing position has been the focus of current studies. According to the systematic review study on the effect of sensory manipulations on postural release changes in individuals with NSLBP, the results are uncertain and further studies are needed. For example, in cases where sensory systems (eg visual, proprioceptive, and vestibular) that are effective in achieving postural control are not manipulated, some studies report greater release size in NSLBP patients, while others find that the size of release is similar to healthy individuals. Sherafat et al. Emphasized that the evaluation of gravity center changes in static environment may be effective in the emergence of these contradictory results. As expressed in this study, standing still on a static platform may be an obstacle to detect small postural stability and balance differences between individuals with and without NSLBP. In this context, testing of geriatric individuals with NSLBP in the standing position on a mobile platform such as the Biodex Balance System (BBS) (Biodex Medical Systems, Shirley, NY) and exposure to more stringent equilibrium conditions will yield more sensitive results in assessing postural stability and balance.

BBS is a device used for objective evaluation of static and dynamic balance, allowing free movement in mediolateral and anteroposterior directions. The validity-reliability studies of the BBS were conducted in various populations including active, non-active, young adult and geriatric individuals, and individuals with ankle sprains. The validity-reliability study of individuals with NSLBP was reported by Sherafat et al. has a strong-excellent correlation with four-square step test, timed-up-and-go test, Berg Balance Scale, and single leg stance test.

Studies have emphasized the use of BBS in geriatric individuals with NSLBP, but no data on the cut-off scores of this system have been found. The determination of a cut-off score with high sensitivity and specificity is thought to be beneficial for detecting deterioration in functional status in geriatric individuals with NSLBP. Therefore, the aim of our study is to determine BBS cut-off scores in geriatric individuals with NSLBP.

ELIGIBILITY:
Inclusion Criteria:

* the presence of episodic low back pain for 12 months or more,
* having a 40 mm pain score on the day of visual analog scale,
* the ability to follow and follow verbal commands,
* to volunteer to participate in the study.

Exclusion Criteria:

* presence of severe spinal pathologies,
* history of spinal surgery,
* presence of neurological deficits,
* diagnosis of any specific low back pain (facet joint problem, disc herniation and sacroiliac joint dysfunction, etc.),
* nerve root compression,
* scoliosis, lordosis or kyphosis,
* cancer or the presence of other autoimmune diseases.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Our study will be planned as a cross-sectional study. 52 geriatric individuals with NSLBP who applied to the Orthopedics and Traumatology Outpatient Clinic will be included in the study if they meet the inclusion criteria. These individuals will be evaluated by an experienced physiotherapist in the laboratory for the variables examined during the day.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Biodex Balance System (BBS) | 6 weeks
  The BBS will be used to assess postural performance of participants. The movable platform of the BBS allows up to 20° of surface tilt in anterior-posterior and medial-lateral directions. The device is equipped with computer software (Biodex, version 3.1; Biodex Medical Systems). Medial-lateral stability index (MLSI) will be assessed.
Antero-posterior stability index | 6 weeks
  Antero-posterior stability index (APSI) will be assessed.
Overall stability index | 6 weeks
  Overall stability index (OSI) will be assessed.

SECONDARY OUTCOMES:
Berg Balance Scale (BergBS) | 6 weeks
  The Berg Balance Scale (BergBS) will be used as a gold-standard test to measure postural performance of participants. The BergBS is a qualitative measure that assesses postural performance via performing functional activities such as reaching, bending, transferring, and standing that incorporates most components of postural control: sitting and transferring safely between chairs; standing with feet apart, feet together, in single-leg stance, and feet in the tandem Romberg position with eyes-open or eyes-closed; reaching and stooping down to pick something off the floor. Each item is scored along a 5-point scale, ranging from 0 to 4, each grade with well-established criteria. Zero indicates the lowest level of function and 4 the highest level of function. The total score ranges from 0 to 56.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sherafat S, Salavati M, Ebrahimi Takamjani I, Akhbari B, Mohammadirad S, Mazaheri M, Negahban H. Intrasession and intersession reliability of postural control in participants with and without nonspecific low back pain using the Biodex Balance System. J Manipulative Physiol Ther. 2013 Feb;36(2):111-8. doi: 10.1016/j.jmpt.2012.12.005. PMID 23499146
- [Result] Dawson N, Dzurino D, Karleskint M, Tucker J. Examining the reliability, correlation, and validity of commonly used assessment tools to measure balance. Health Sci Rep. 2018 Oct 27;1(12):e98. doi: 10.1002/hsr2.98. eCollection 2018 Dec. PMID 30623052
- [Result] Arifin N, Abu Osman NA, Wan Abas WA. Intrarater test-retest reliability of static and dynamic stability indexes measurement using the Biodex Stability System during unilateral stance. J Appl Biomech. 2014 Apr;30(2):300-4. doi: 10.1123/jab.2013-0130. Epub 2013 Jul 20. PMID 23878204